CLINICAL TRIAL: NCT03392636
Title: Comparison of Recurrence Rate of Ferguson & Gross Herniotomy With Mitchell Banks Herniotomy in Children Older Than 2 Years
Brief Title: Comparison of Recurrence Rate of 2 Herniotomy Techniques in Children Older Than 2 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fatima Numeri, assisstant professor, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 212/RC/KEMU
Record Dates: First submitted 2017-12-08; First posted 2018-01-08 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-03

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: Group A will get Mitchell Banks herniotomy done and Group B will get Fergusson Gross Herniotomy done.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Mitchell Banks Herniotomy
  Interventions: Procedure: Herniotomy
- Group B (Experimental): Fergusson Gross Herniotomy
  Interventions: Procedure: Herniotomy

INTERVENTIONS:
Procedure: Herniotomy — In Mitchell Banks Herniotomy, one of investigators will do herniotomy without opening inguinal canal and in Ferguson Gross Herniotomy , one of investigators will do herniotmy by opening inguinal canal.
  Other Names: Mitchell Banks Herniotomy; Fergusson Gross Herniotomy

SUMMARY:
the study is basically aimed at comparing two techniques of herniotomy by comparing there recurrence rates

DETAILED DESCRIPTION:
in this study, the principal investigator will operate upon patients aged between 2 years and 12 years by two techniques. in technique called mitchell banks technique, inguinal canal will not be opened and in Fergusson gross technique, it will be opened

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients of either gender above age of 2 years and below 14 years of age presenting in pediatric surgery Mayo hospital lahore

Exclusion Criteria:

* sliding hernia strangulated hernia pts with connective tissue disorders pts with undesccended testis patients with hydrocele hernia with internal ring 2cm or more in size

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
recurrence | 6 months
  Recurrence will be assessed 6 months after the procedure

SECONDARY OUTCOMES:
size of incision | upto 6 months, will be noted at the end of every procedure
  length of incision will be noted
operation time | upto 6 months, will be noted at the end of every procedure
  total operative time will be noted
Intra operative complications | upto 6 months, will be noted at the end of every procedure
  Tearing of processus vaginalis, ilioinguinal nerve injury
post-operative complications | will be noted on follow up at 7 days post op
  Wound Infection b. Scrotal Edema c. Haematoma d. TesticularRetraction
Testicular Atrophy | 6 months after procedure
  testicular atrophy will be noted

CONTACTS AND LOCATIONS:
Locations (1):
- KEMU, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2016-11-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT03392636/ICF_000.pdf